CLINICAL TRIAL: NCT03487978
Title: The Migrainous Brain: a Prospective Research for Longitudinal Changes of Brain Networks in Migraine
Brief Title: Longitudinal Changes of Brain Functional Connectivity in Migraine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: National Research Foundation of Korea (Other); Sungkyunkwan University (Other)
Responsible Party: Principal Investigator, Chin-Sang Chung, MD, PhD, Professor of neurology, Samsung Medical Center
Other Study IDs: 2017-03-113
Record Dates: First submitted 2018-03-27; First posted 2018-04-04 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraineurs: Patients diagnosed with migraine based on the ICHD-3 beta will undergo 3-tesla resting-state functional MRI.
  Interventions: Diagnostic Test: resting-state functional MRI
- Control: Normal controls without headaches will undergo 3-tesla resting-state functional MRI.
  Interventions: Diagnostic Test: resting-state functional MRI

INTERVENTIONS:
Diagnostic Test: resting-state functional MRI — 1. To ensure inter-ictal fMRI, confirm that the subject has no migraine for at least 48 hours before the procedure.
  2. Record the time difference between the date on the day of fMRI and the date of the last headache attack and record whether the headache on the day of fMRI is absent or not.
  3. On the third day after MRI, examine whether the subject has headache or not.

SUMMARY:
The purpose of this study is to identify a core fMRI feature that determines migrainous brain and plastic fMRI features that changes with longitudinal courses of migraine.

DETAILED DESCRIPTION:
Migraine is associated with functional alterations in specific brain networks. The investigators aimed to identify network abnormalities which remain unchanged throughout the longitudinal course of migraine. The investigators also aimed to identify networks which change in association with changes in migraine frequency and associated psychiatric conditions. The investigators expect these can serve as neuroimaging biomarkers for diagnosis of migraine brain and monitoring of disease severity.

ELIGIBILITY:
Inclusion Criteria:

Migrainuers :

1. age 18-50 years
2. migraine with or without aura as defined by the third edition of the International Classification of Headache Disorders (ICHD-3 beta)
3. if female, before the onset of menopausal

Controls:

1. age 18-50 years
2. no headache disorder other than Infrequent episodic tension-type headache as defined by the ICHD-3 beta

Exclusion criteria:

1. contraindicated to MRI
2. pregnancy
3. require sedation treatment because of claustrophobia when performing MRI
4. predicted to be unable to write the headache diary due to cognitive decline
5. refuse study procedure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Controls and migraineurs who visited to a single university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Core fMRI features for migraine brain | 1-year follow-up (2nd year)
  Among significant networks identified by ICA, we will identify altered networks which remain unchanged in follow-up resting-state fMRI in 1 year.

SECONDARY OUTCOMES:
Candidate fMRI features for migraine | Baseline (1st year)
  Using baseline resting-state fMRI, altered brain networks associated with migraine will be identified by independent component analysis (ICA) between patients and controls.
Dynamic fMRI features for disease severity | 1-year follow-up (2nd year)
  Among significant networks identified by ICA, we will identify altered networks which change in association with changes in headache frequency in follow-up resting-state fMRI in 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Ji Lee, MD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea